CLINICAL TRIAL: NCT01057524
Title: The Use of High Frequency Chest Wall Oscillation During an Acute Infective Pulmonary Exacerbation of Cystic Fibrosis
Brief Title: High Frequency Chest Wall Oscillation and Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0708/10
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2012-02

CONDITIONS: Cystic Fibrosis
Keywords: Airway clearance; Cystic fibrosis; High frequency chest wall oscillation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Chest Wall Oscillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Airway Clearance Technique (Active Comparator): Two self administered treatment sessions a day and two treatments a day assisted by a Physiotherapist both using the patient's usual airway clearance method.
  Interventions: Other: Usual airway clearance
- High Frequency Chest Wall Oscillation (HFCWO) (Experimental): Two self administered treatments a day using HFCWO and two treatment sessions a day assisted by a Physiotherapist using their 'usual' airway clearance method.
  Interventions: Device: High Frequency Chest Wall Oscillation (HFCWO)

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillation (HFCWO) — Airway clearance using the high frequency chest wall oscillator device
  Other Names: 'The Vest', Hill Rom Model 205
  Arms: High Frequency Chest Wall Oscillation (HFCWO)
Other: Usual airway clearance — Airway clearance treatments using the active cycle of breathing techniques, autogenic drainage, positive expiratory pressure, manual techniques or oscillating positive expiratory pressure
  Other Names: Airway clearance techniques (ACT's)
  Arms: Usual Airway Clearance Technique

SUMMARY:
High frequency chest wall oscillation (HFCWO) has been shown to increase tracheal mucus clearance compared with a control group. These observations led to the development of The Vest® which is a non-stretchable jacket connected to an air-pulse generator and worn by the patient over the chest wall. The generator rapidly inflates and deflates The Vest®, which gently compresses and releases the chest wall between 5 and 20 times per second. This generates mini-coughs that are said to dislodge mucus from the bronchial walls and to facilitate its movement up the airways. The Vest® has been shown to reduce the viscosity of mucus and this should further enhance mucus clearance.

People with cystic fibrosis (CF), admitted to hospital with an acute infective pulmonary exacerbation, should increase the frequency and duration of their airway clearance sessions owing to the increase in quantity and viscosity of purulent bronchial secretions.In the United Kingdom, and in many other countries, the availability of physiotherapists to assist with the recommended number of daily treatments is insufficient to meet patient need. If the use of high frequency chest wall oscillation, in addition to 'usual' self airway clearance techniques, in the early morning and evening was to facilitate recovery from an exacerbation, this would indicate an important place for high frequency chest wall oscillation in the management of people with cystic fibrosis.

Hypothesis:

The addition of high frequency chest wall oscillation to twice daily supervised physiotherapy is as effective as the addition of self treatment in facilitating recovery from an acute infective pulmonary exacerbation, as measured by improvement in lung function, specifically forced expiratory volume in one second (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Hospitalised patients admitted with a pulmonary infection
* Forced expiratory volume in one second (FEV1)of 15% predicted or over
* 16 years of age or over

Exclusion Criteria:

* Current severe haemoptysis
* Rib fractures or history of spontaneous rib fractures
* pregnancy
* Lung abscess
* End stage disease
* Requiring more than two assisted treatment sessions per day
* Requiring treatment with positive pressure
* Inability to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in forced expiratory volume in one second (FEV1) | 7days

SECONDARY OUTCOMES:
Wet weight of sputum expectorated | 24 hours
Length of time to next course of intravenous antibiotics | Within 6 monthsof completing study
Rate of change of C-reactive protein | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hodson, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Burnham P, Stanford G, Stewart R. Autogenic drainage for airway clearance in cystic fibrosis. Cochrane Database Syst Rev. 2021 Dec 15;12(12):CD009595. doi: 10.1002/14651858.CD009595.pub3. PMID 34910295